CLINICAL TRIAL: NCT04193761
Title: COMPARISON BETWEEN SERUM TAURINE AND SPECIFIC TUMOR MARKERS FOR EARLY DETECTION AND DIAGNOSIS OF HCC IN EGYPTIAN PATIENTS
Brief Title: TAURINE and HCC PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HAM00077
Record Dates: First submitted 2019-12-07; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Taurine in HCC

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator)
  Interventions: Diagnostic Test: taurine level
- Chronic hepatitis (Active Comparator)
  Interventions: Diagnostic Test: taurine level
- Cirrhosis (Active Comparator)
  Interventions: Diagnostic Test: taurine level
- Hepatocellular carcinoma (Active Comparator)
  Interventions: Diagnostic Test: taurine level

INTERVENTIONS:
Diagnostic Test: taurine level — Taurine: determined by High-Performance Liquid Chromatography according to the pre-column extraction and derivatization methodology of McMahon et al. in the present work we use the Shimadzu, Japan HPLC model LC-10 AT.

SUMMARY:
Serum taurine level beside (AFP and AFU) are of great value in early diagnosis in HCC Egyptian patients and may have a rule in identifying end-stage liver disease (ESLD) patients candidate for LDLT.

DETAILED DESCRIPTION:
Taurine has been demonstrated to have a direct and indirect antioxidant effect and to display antineoplastic activity by preventing angiogenesis and enhancing tumor cell apoptosis. Also it was suggested that measurement of serum taurine level in hepatic patients beside fibroscan is of great value in the early diagnosis of any fibrotic and cancerous liver changes.Aim of the work was to correlate serum taurine level with the levels of the specific tumor markers (α- fetoprotein and α-L-fucosidase ) for early diagnosis of different stages of HCC in Egyptian patients.

This observational case-control study was conducted in the Tropical Medicine Department, Ahmed Maher Teaching Hospital. Eighty hepatic patients were assigned to three groups (Chronic hepatitis, Cirrhosis and HCC). Twenty healthy subjects were enrolled as a control group. Serum levels of AFP, AFU, and taurine beside complete biochemical analysis and liver biopsies from all selected patients were done. Patients who accepted to be a candidate for living donor liver transplant (LDLT) were referred to Ain Shams University Specialized Hospital (ASUSH) liver transplant unit.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis
* Cirrhosis
* HCC patients

Exclusion Criteria:

* Patient refusal
* Bleeding tendency
* Tense ascites
* Inability to obtain a liver biopsy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Taurine level among patients groups | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: No